CLINICAL TRIAL: NCT05236842
Title: Efficacy, Safety and Tolerability of Three Doses of Sulthiame in Patients With Obstructive Sleep Apnea.
Brief Title: Efficacy, Safety and Tolerability of Sulthiame in Patients With Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STM-042/K; 2021-002926-26 (EudraCT Number)
Record Dates: First submitted 2022-01-20; First posted 2022-02-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: sulthiame; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — sulthiame

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sulthiame 100 mg (Active Comparator): Sulthiame film-coated tablets 100 mg once daily 15 weeks
  Interventions: Drug: Sulthiame
- Sulthiame 200 mg (Active Comparator): Sulthiame film-coated tablets 200 mg once daily 15 weeks
  Interventions: Drug: Sulthiame
- Sulthiame 300 mg (Active Comparator): Sulthiame film-coated tablets 300 mg once daily 15 weeks
  Interventions: Drug: Sulthiame
- Placebo (Placebo Comparator): Placebo film-coated tablets once daily 15 weeks
  Interventions: Drug: Sulthiame

INTERVENTIONS:
Drug: Sulthiame — oral
  Other Names: Ospolot

SUMMARY:
multi-center, randomized, double-blind, placebo-controlled, dose-finding, 4-arm, parallel assignment study to evaluate the efficacy of three different doses of sulthiame (STM) compared to placebo on sleep apnea activity in adult patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Primary objective: To evaluate the efficacy of 3 different doses of Sulthiame (STM) compared to placebo on sleep apnea activity in adult patients with moderate to severe obstructive sleep apnea (OSA) after at least 12 weeks of treatment at target dose

Secondary objectives: To evaluate the effect of 3 different doses of STM after at least 12 weeks of treatment at target dose in patients with moderate to severe OSA on apnea/hypopnea events, hypoxic burden, sleep quality, daytime sleepiness, patient's perception of symptoms and well-being, comorbidity-related outcomes and safety and tolerability of STM

Exploratory objective: To evaluate potential predictive biomarker (eg, blood gas analysis parameters or additional polysomnography [PSG] variables) with regard to efficacy

ELIGIBILITY:
Key Inclusion Criteria:

* OSA diagnosis according to the International Classification of Sleep Disorders - Third Edition criteria with an AHI of ≥15 documented by PSG or polygraphy (PG).
* Currently not treated with continuous positive airway pressure (CPAP) or mandibular advancement device (MAD) due to patient-reported:
* non-tolerability; and/or
* non-compliance; and/or
* not willing to use CPAP or MAD (treatment-naïve patients)

Key Exclusion Criteria:

* Any OSA treatment within the last 4 weeks prior to screening
* Fulfill criteria for a dominant central sleep apnea syndrome or dominant Cheyne Stokes respiration
* Other clinically significant sleep disorder including periodic limb movement disorder, restless leg syndrome, periodic limb movement arousal index (PLMAI) of >15*, insomnia, parasomnia or narcolepsy

  * as part of PSG baseline assessment
* Hypoventilation or hypoxemia due to chronic obstructive pulmonary disease or other respiratory condition
* Clinically relevant craniofacial malformation
* Any upper airway surgery for OSA within the last 12 months prior to baseline
* Patients who underwent an obesity surgery within the last 2 years prior to baseline or patients actively participating in any weight loss treatment program or use of any weight loss medication (prescription or over-the-counter) within 1 month prior to the first PSG night.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Relative change in apnea-hypopnea index (AHI) from baseline to Week 15 (at least 12 weeks of treatment at target dose) measured by PSG | from baseline to week 15
  change in apnea-hypopnea index (AHI)

SECONDARY OUTCOMES:
Number and percentage of patients reporting adverse events, treatment-emergent adverse events (TEAEs) , serious TEAEs, related TEAEs, related serious TEAEs, TEAEs leading to discontinuation of study drug. | from baseline to week 15
  Two-sided 95% confidence intervals for the difference in patient incidence between each sulthiame treatment group and placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumocare SRL, Namur, Belgium

REFERENCES:
- [Derived] Randerath W, Grote L, Stenlof K, Fietze I, Chevts J, Buntinx E, Albares J, Kuhn K, Hansen C, Volp A, Hedner J; FLOW study investigators. Sultiame once per day in obstructive sleep apnoea (FLOW): a multicentre, randomised, double-blind, placebo-controlled, dose-finding, phase 2 trial. Lancet. 2025 Oct 25;406(10514):1983-1992. doi: 10.1016/S0140-6736(25)01196-1. Epub 2025 Oct 9. PMID 41077049